CLINICAL TRIAL: NCT00246454
Title: Circadian Rhythms and Sleep in Familial Delayed Sleep Phase Syndrome (DSPS) and Advanced Sleep Phase Syndrome (ASPS)
Brief Title: Circadian Rhythms and Sleep in Familial DSPS and ASPS
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Phyllis Zee, Benjamin and Virginia T. Boshes Professor of Neurology, Northwestern University
Other Study IDs: 341; R01HL069988 (NIH)
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Circadian Rhythm Sleep Disorder
Keywords: circadian; advanced sleep phase; delayed sleep phase
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: People with delayed sleep phase syndrome (DSPS).
- 2: People with advanced sleep phase syndrome (ASPS).
- 3: Control group (people with intermediate sleep patterns).

SUMMARY:
The purpose of this study is to determine the properties of circadian rhythms and sleep propensity in familial advanced and delayed sleep phase syndrome (DSPS).

DETAILED DESCRIPTION:
BACKGROUND:

Tremendous progress in the past few years has led to the identification of several circadian clock genes. This now makes it possible to determine how alterations of human circadian clock genes and their expression could lead to differences in circadian and sleep/wake cycle phenotypes. Of particular interest for understanding genetics of the human circadian system are individuals with sleep phase disorders, such as DSPS and advanced sleep phase syndrome (ASPS), because recent studies indicate a genetic basis for these disorders. While it is assumed that both ASPS and DSPS are disorders of circadian timing, little is known about how the circadian clock system, or its interaction with sleep processes, are affected in these individuals.

DESIGN NARRATIVE:

Participants will complete questionnaires and actigraphy to determine sleep patterns and quality.

ELIGIBILITY:
Inclusion Criteria for ASPS Participants:

* Morning type score on the Horne-Ostberg questionnaire
* Advanced melatonin onset

Inclusion Criteria for DSPS Participants:

* Evening type score on the Horne-Ostberg questionnaire
* Delayed melatonin onset

Inclusion Criteria for Controls:

* A stable sleep/wake pattern with a normal phase relationship to the environment and no history of sleep disorders

Exclusion Criteria for all subjects:

* Sleep disorder, other than DSPS or ASPS, as assessed by the Pittsburgh Sleep Quality Index and/or by polysomnogram
* History of cognitive or other neurological disorders
* History of Diagnostic and Statistical Manual-IV criteria for any major psychiatric disorder, alcohol or substance abuse
* Abnormal mood as assessed by the Hamilton Depression Scale
* History of, or concurrent, unstable or serious medical illness
* Current use of psychoactive medications, including antidepressants, anxiolytics, neuroleptics, anticonvulsants, hypnotics, and stimulant medications
* Shift work
* Having a daily caffeine intake greater than 4 cups per day
* Smoking
* Travel across more than 2 time zones within 90 days of the study
* Pregnancy or the desire to become pregnant during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with circadian rhythm sleep disorders and healthy age and gender matched controls
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2003-09; Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Sleep | 1 night
  Assessment of sleep parameters

SECONDARY OUTCOMES:
Circadian Timing | 3 days
  Assessment of circadian activity profiles

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis C. Zee, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reid K. J., Zee P.C. (2005) Circadian Disorders of the Sleep-Wake Cycle. Kryger, Roth, Dement (ed's) Principle and Practices of Sleep Medicine, 4th Ed. Saunders.
- [Result] Baron KG, Reid KJ, Kern AS, Zee PC. Role of sleep timing in caloric intake and BMI. Obesity (Silver Spring). 2011 Jul;19(7):1374-81. doi: 10.1038/oby.2011.100. Epub 2011 Apr 28. PMID 21527892
- [Result] Reid KJ, Jaksa AA, Eisengart JB, Baron KG, Lu B, Kane P, Kang J, Zee PC. Systematic evaluation of Axis-I DSM diagnoses in delayed sleep phase disorder and evening-type circadian preference. Sleep Med. 2012 Oct;13(9):1171-7. doi: 10.1016/j.sleep.2012.06.024. Epub 2012 Aug 19. PMID 22910327
- [Result] Baron KG, Reid KJ, Horn LV, Zee PC. Contribution of evening macronutrient intake to total caloric intake and body mass index. Appetite. 2013 Jan;60(1):246-251. doi: 10.1016/j.appet.2012.09.026. Epub 2012 Oct 2. PMID 23036285
- [Result] Reid KJ, Santostasi G, Baron KG, Wilson J, Kang J, Zee PC. Timing and intensity of light correlate with body weight in adults. PLoS One. 2014 Apr 2;9(4):e92251. doi: 10.1371/journal.pone.0092251. eCollection 2014. PMID 24694994
- [Result] Wilson J 4th, Reid KJ, Braun RI, Abbott SM, Zee PC. Habitual light exposure relative to circadian timing in delayed sleep-wake phase disorder. Sleep. 2018 Nov 1;41(11):zsy166. doi: 10.1093/sleep/zsy166. PMID 30423177
- [Result] Joo EY, Abbott SM, Reid KJ, Wu D, Kang J, Wilson J, Zee PC. Timing of light exposure and activity in adults with delayed sleep-wake phase disorder. Sleep Med. 2017 Apr;32:259-265. doi: 10.1016/j.sleep.2016.09.009. Epub 2016 Nov 9. PMID 27964860